CLINICAL TRIAL: NCT00418626
Title: A Phase I, Single Center, Open-label, Single Oral Dose, Study to Assess the Pharmacokinetics of Nilotinib in Subjects With Impaired Hepatic Function and Healthy Subjects With Normal Hepatic Function
Brief Title: Pharmacokinetics of Nilotinib in Subjects With Impaired Hepatic Function and Healthy Subjects With Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107A2116
Record Dates: First submitted 2007-01-03; First posted 2007-01-05 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
Keywords: nilotinib; hepatic impairment; Child-Pugh scale; PK; healthy, subject(s); Subjects with impaired hepatic function and healthy subjects
MeSH Terms: interventions — nilotinib

ARMS (1):
- Nilotinib (Experimental)
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib
  Other Names: AMN107

SUMMARY:
This study will be a formal assessment of the impact of hepatic function impairment on the pharmacokinetics of nilotinib

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male (18 -70 yrs)
2. Body weight must be ≥ 50 kg and < 120 kg, with a body mass index (BMI) >18 but < 35.
3. Laboratory parameters values within the normal range

Exclusion Criteria:

1. Contraindication or hypersensitivity to receiving nilotinib
2. Smokers or those who use of tobacco products or products containing nicotine
3. A past medical history of clinically significant Electrocardiogram abnormalities or a history/family history of long QT-interval syndrome.
4. History of fainting spells.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-11; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of nilotinib

SECONDARY OUTCOMES:
impact on hepatic function assessed by laboratory values and an electrocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (1):
- Richmond, Virginia, United States

REFERENCES:
- [Derived] Yin OQ, Gallagher N, Tanaka C, Fisher D, Sethuraman V, Zhou W, Lin TH, Heuman D, Schran H. Effects of hepatic impairment on the pharmacokinetics of nilotinib: an open-label, single-dose, parallel-group study. Clin Ther. 2009;31 Pt 2:2459-69. doi: 10.1016/j.clinthera.2009.11.015. PMID 20110053